CLINICAL TRIAL: NCT06912815
Title: Comparative Analysis of Curative Effect Ustekinumab Combined With Semi Enteral Nutrition and Exclusive Enteral Nutrition in Preoperative Optimization of Crohn's Disease: A Multicenter, Prospective, Randomized, Controlled Study
Brief Title: Ustekinumab With Semi-EN vs Exclusive EN for Preoperative Crohn's Disease Optimization.
Acronym: USE-OPT CD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiang Gao (Other)
Responsible Party: Sponsor-Investigator, Xiang Gao, Director of Gastroenterology, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-069
Record Dates: First submitted 2025-03-24; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease (CD)
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ustekinumab and semi enteral nutrition (Experimental)
  Interventions: Biological: ustekinumab and semi enteral nutrition
- Exclusive enteral nutrition (Experimental)
  Interventions: Other: Exclusive enteral nutrition

INTERVENTIONS:
Biological: ustekinumab and semi enteral nutrition — Preoperative treatment optimization involves a single intravenous induction with UST, followed by 6 weeks of oral/nasal feeding with semi-enteral nutrition.
  Arms: ustekinumab and semi enteral nutrition
Other: Exclusive enteral nutrition — Preoperative optimized treatment with 6 weeks of oral/nasal feeding of exclusive enteral nutrition alone.
  Arms: Exclusive enteral nutrition

SUMMARY:
Ustekinumab (UST) is a novel biologic agent that targets and binds to Interleukin-12 (IL-12) and Interleukin-23 (IL-23), and is approved for inducing and maintaining remission in Crohn Disease(CD). Currently, it is believed that the use of UST for the preoperative treatment of CD patients is generally safe and does not increase surgical complications, and it can be used for preoperative treatment of CD. However, there is still a lack of literature reporting the role of UST in preoperative optimization for CD. Semi-enteral nutrition refers to the provision of more than 50% of the energy required by the human body through enteral nutrition preparations. Semi-enteral nutrition can improve the nutritional status of patients with CD, but it does not induce remission of active disease. The treatment method of UST combined with semi-enteral nutrition can not only induce disease remission, but also improve the nutritional status of patients. Therefore, can the combined treatment regimen replace Exclusive Enteral nutrition (EEN) as a new therapy for preoperative optimization of CD? At present, there is a lack of relevant research, so this study intends to conduct a multi-center, prospective, randomized controlled trial to compare the efficacy differences between UST+semi-enteral nutrition and EEN in preoperative optimization for CD, and to clarify the preoperative optimization effect of UST combined with semi-enteral nutrition therapy.

ELIGIBILITY:
Inclusion Criteria:

* CD patients with surgical indications, who are scheduled for partial intestinal resection and anastomosis;
* CD patients diagnosed prior to surgery;
* Patients aged 18-65;
* CDAI score of >150;
* For patients with peritoneal abscess, they must receive adequate antibiotics and drainage prior to enrollment, and be confirmed to be free of infection before enrolling in the study;
* The patients agree to participate in the study and sign an informed consent form;
* Patients who have not used ustekinumab prior to surgery;
* Patients who have tried other treatments and found them ineffective, and plan to stop using them and schedule surgery.

Exclusion Criteria:

* Emergency surgery;
* Had received exclusive enteral nutrition support within 3 months prior to surgery;
* Unable to tolerate enteral nutrition;
* Failed with UST;
* Pregnant or with co-existing intestinal outside organ dysfunction, tumor, rheumatological or immunological diseases, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Preoperative clinical remission rate | From enrollment to the end of treatment at 6 weeks
  Patients enrolled should collect basic information such as height, weight, disease activity at baseline, and complete examinations including complete blood count, blood biochemistry (electrolytes, liver and kidney function), C-reactive protein, CTE/MRE, intestinal color Doppler ultrasound, nutritional risk NRS2002 score, colonoscopy, as well as iron, calcium, folic acid, and other trace elements. These indicators should be rechecked after 6 weeks post-enrollment.Compare the clinical remission rates of two groups of patients after treatment.

SECONDARY OUTCOMES:
Incidence of complications within 30 days post-surgery | Within 30 days post-surgery
  Postoperative day 3: Complete the QoR-15 questionnaire; Postoperative day 7: Re-examine blood routine, liver and kidney function, CRP, and intestinal color Doppler ultrasound; Postoperative week 4: Re-examine blood routine, liver and kidney function, CRP, intestinal color Doppler ultrasound, and complete the IBDQ questionnaire.
Changes in nutritional and inflammatory indicators before and after optimization | From enrollment to the end of treatment at 6 weeks
  Compare the baseline and the height, weight, and inflammatory indicators (including complete blood count, CRP, liver function, etc.) of two groups of patients after 6 weeks of treatment.
Surgical anastomosis rate for phase I | From enrollment to the end of surgery
  Compare the anastomosis rate after the first stage of surgery between two groups of optimized patients.
Clinical recurrence rate at 12 weeks post-operation | Within 12 weeks post-surgery
  Clinical relapse: Patients in clinical remission who, at any visit, have a Crohn's Disease Activity Index (CDAI) of 150 or higher.
Histological status of surgical margins | From enrollment to the end of surgery
  Comparing the histological conditions of surgical margins in patients after optimization treatment between two groups, to verify whether UST + semi-enteral nutrition has a better therapeutic effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided